CLINICAL TRIAL: NCT04839575
Title: Prospective, Double-Blind, Placebo-Controlled, Crossover Study of the Efficacy and Safety of Latiglutenase Treatment in Type 1 Diabetes Patients With Celiac Disease While Undergoing Periodic Gluten Exposure
Brief Title: Study of Latiglutenase in T1D/CD Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid-19 interruptions and enrollment challenges
Sponsor: Entero Therapeutics (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Immunogenics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IMGX003-NIDDK-1921; 1R44DK121606-01 (NIH)
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2023-07

CONDITIONS: Celiac Disease
Keywords: Celiac
MeSH Terms: conditions — Celiac Disease | interventions — ALV003

STUDY DESIGN:
Intervention Model Description: A two-period crossover design will be used where the treatment sequences will be assigned at random.
Who Masked: Participant, Investigator
Masking Description: The PI, CRA and study biostatistician will be masked until database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Latiglutenase (Active Comparator): IMGX003
  Interventions: Drug: Latiglutenase
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Latiglutenase — Administered orally (daily)
  Other Names: IMGX003
  Arms: Latiglutenase
Drug: Placebo — Administered orally (daily)
  Arms: Placebo

SUMMARY:
This is a phase 2, single-center prospective, double-blind, placebo-controlled, crossover study in Type 1 diabetes and celiac disease subjects attempting a GFD for at least one year prior to screening.

DETAILED DESCRIPTION:
This is a phase 2, single-center prospective, double-blind, placebo-controlled, crossover study in Type 1 diabetes and celiac disease subjects attempting a GFD for at least one year prior to screening. Seropositive subjects (blood test confirmed at Visit 0) will be scheduled for a Screening Visit (Visit 1) whereas seronegative subjects will be discontinued from study participation (screen failures). Subjects who meet Visit 1 protocol enrollment criteria will be enrolled.

ELIGIBILITY:
Inclusion Criteria (select):

* Confirmed CD diagnosis
* Confirmed T1D diagnosis
* Seropositive
* Gluten free diet (12 months minimum)
* Experienced at least one self-reported moderate or greater severity symptom during the last 28 day period
* Willing to take study treatment daily
* Must sign informed consent

Exclusion Criteria (select):

* Wheat allergy
* History of peptic ulcer disease, esophagitis, IBS, IBD
* Active colitis
* Subjects with known rapid gastric emptying (post-bariatric surgery, Billroth I or II surgery)
* Chronic infectious gastrointestinal illness or acute infectious gastrointestinal illness within the 4 week period prior to screening
* Known refractory celiac disease (RCD1 or RCD2)
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Symptom Severity Reduction | 6 months
  The primary efficacy endpoint of this study is absolute mean reduction in symptom severity relative to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: David Maahs, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No